CLINICAL TRIAL: NCT02056808
Title: SMT C1100 - A Phase 1b, Open-label, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Paediatric Patients With Duchenne Muscular Dystrophy
Brief Title: A Phase 1b Study of SMT C1100 in Subjects With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMT C11002
Record Dates: First submitted 2013-11-21; First posted 2014-02-06 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — SMT C1100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SMT C1100 (Experimental): Patients will be studied in 3 groups (Groups A to C), with each group consisting of 4 patients aged between 5 to 11 years. It is planned that doses for Groups A to C will be administered in an escalating manner after safety review for each dose group.
  Interventions: Drug: SMT C1100

INTERVENTIONS:
Drug: SMT C1100 — Comparison of safety and pharmacokinetic of different dosages of drug

SUMMARY:
The purpose of this study is to determine whether increasing doses of SMT C1100 are safe, well tolerated and achieve appropriate blood levels in patients with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
Primary Objective: To determine the safety and tolerability of single and multiple oral doses of SMT C1100 in patients with Duchenne Muscular Dystrophy (DMD).

Secondary Objectives: To determine the single and multiple oral dose pharmacokinetics of SMT C1100 and its metabolites in patients with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be males of any ethnic origin with a genetic diagnosis of DMD.
* Children between 5 and 11 years of age.
* A parent/legal guardian must date and sign a written consent on behalf of the patient, according to International Conference on Harmonisation (ICH) and local regulations. This person must understand the contents of the consent, requirements of the study and have had an opportunity to review questions with a medically trained member of the site study team.
* The patient is willing to give verbal or written age appropriate assent to participate.
* For safety reasons, the patient's parent/legal guardian must have a good understanding of the English language, as this is the only language the consent/assent forms are written in, and understand the requirements for reporting of any adverse event to the Investigator.

Exclusion Criteria:

* Enrollment or participation in any therapeutic clinical trial within the prior 3 months or 5 times the half-life (whichever is longer).
* Initiation or change (other than dose modifications for body weight) of systemic corticosteroid therapy within 2 months prior to the start of dose administration or discontinuation of corticosteroids within 30 days prior to the start of dose administration.
* Known hypersensitivity to the excipients of the study drug or a previous history of drug allergy.
* Use of the following therapies is prohibited during the study and for at least 5 half-lives prior to the start of dose administration: Inducers of cytochrome P450 CYP1A2 (eg, carbamazepine, phenytoin, primidone, rifampin, omeprazole, and barbiturates), and moderate and strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin, enoxacin, mexiletine; propafenone, zileuton). Substrates of CYP1A2 with narrow therapeutic windows (e.g., tacrine, theophylline, methadone, mexiletine). Nicotine, including exposure to daily passive smoking to minimize cytochrome P450 CYP 1A induction. Chargrilled food, cruciferous vegetables, caffeine, tea, and any xanthine containing foods, and drinks are prohibited from 36 hours prior to check-in until final discharge from study. Herbal supplements and homeopathic preparations (unless approved by medical monitor).
* Need for mechanical ventilation.
* Non ambulatory.
* Any clinically significant acute illness within 4 weeks of the start of dose administration.
* Any co-morbidity that, in the opinion of the Investigator, increases the risk of participating in the study.
* Symptomatic cardiomyopathy that in the opinion of the Investigator prohibits participation in this study.
* Abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study.
* Any clinically significant medical condition, other than DMD that in the opinion of the Investigator may increase the risk of participating in the study or interfere with the interpretation of safety or efficacy evaluations (e.g., concomitant illness, psychiatric condition or behavioral disorder).
* Exposure to daily passive smoking (including parent/legal guardian, siblings) so as to minimize environmental factors causing cytochrome P450 CYP 1A induction. For information SMT C1100 is metabolized by cytochrome P450 CYP 1A.
* Excessive exercise (Investigator opinion).

Ages: 5 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | After 10 days of treatment phase
  To determine the safety and tolerability of single and multiple oral doses of SMT C1100 in patients with Duchenne Muscular Dystrophy (DMD) by assessing the participants adverse events, ECG results, vital signs and laboratory tests.

SECONDARY OUTCOMES:
Pharmacokinetic parameters at different dose levels | After single oral dose and after 10 days of treatment phase
  Plasma concentration of SMT C1100 calculated at each time point for each subject (sample size (n), mean, standard deviation (SD), percentage of coefficient of variation (%CV), geometric mean, median, minimum, and maximum for the parent and the major metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Spinty, MD, Principal Investigator — Alder Hey Children's NHS Foundation Trust; Helen Roper, MD, Principal Investigator — Heart of England NHS Foundation Trust - Heartlands Hospital; Imelda Hughes, MD, Principal Investigator — Central Manchester University Hospitals NHS Foundation Trust - Royal Manchester Childrens Hospital; Franceso Muntoni, MD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Heart of England NHS Foundation Trust - Heart Lands Hospital, Birmingham
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street for Children NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust- Royal Manchester Children's Hospital, Manchester